CLINICAL TRIAL: NCT06817096
Title: Phase 3, Multicenter, Parallel, Randomized, Single-blind, Placebo-controlled Clinical Trial to Evaluate the Efficacy and Safety of Nitazoxanide 600 Mg Administered Twice Daily, in the Outpatient Treatment of COVID-19 and Influenza
Brief Title: Efficacy and Safety of Nitazoxanide 600 Mg in the Outpatient Treatment of COVID-19 and Influenza
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Azidus Brasil (Industry)
Collaborators: Farmoquimica S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FQMNita
Record Dates: First submitted 2025-02-06; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Covid 19; Influenza
Keywords: nitazoxanide; outpatient treatment
MeSH Terms: conditions — COVID-19; Influenza, Human | interventions — nitazoxanide; Tablets

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- placebo (Placebo Comparator): take placebo orally, twice daily for 7 days.
  Interventions: Drug: Nitazoxanide 600Mg Oral Tablet / placebo oral tablet
- nitazoxanide (Experimental): take nitazoxanide 600 mg orally, twice daily for 7 days
  Interventions: Drug: Nitazoxanide 600Mg Oral Tablet / placebo oral tablet

INTERVENTIONS:
Drug: Nitazoxanide 600Mg Oral Tablet / placebo oral tablet — 1 tablet every 12 hours

SUMMARY:
2. Participants will:

* Take nitazoxanide 600mg (or placebo) orally twice daily for 7 days, for a total of 14 doses.
* Visit the clinic on the 7th day of treatment for a check-up and safety tests.
* Keep a diary of their symptoms and other medications used

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form;
* Male or female;
* Age ≥ 18 years;
* COVID-19 or influenza diagnosed by rapid test, with symptom onset less than 48 hours ago;
* Clinical condition compatible with outpatient treatment.

Exclusion Criteria:

* Known hypersensitivity to nitazoxanide;
* History of cardiomyopathies, hepatopathies, or nephropathies;
* Antineoplastic treatment with chemotherapy or radiotherapy;
* Severe autoimmune diseases with immunosuppression;
* Transplant recipients;
* Any uncompensated systemic disease at the investigator's discretion;
* Participation in clinical studies in the last 12 months;
* Pregnant or breastfeeding individuals;
* Suspected bacterial coinfection or prescription of antibiotic therapy at enrollment;
* Diagnosis of neurological disease (traumatic brain injury, stroke, Parkinson's disease, Alzheimer's disease, other dementias);
* Diagnosis of developmental disorder (ADHD, ASD, learning disabilities, intellectual disability, Rett syndrome);
* Significant hearing or vision impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the Effectiveness of Nitazoxanide in the Outpatient Treatment of COVID-19 | From enrollment to the end of treatment will last up to 60 days
  The evaluation will be conducted by comparing the nitazoxanide and placebo groups regarding the time to symptom resolution (fever, cough, runny nose, nasal congestion, sore throat, fatigue, headache, muscle pain, sweating, or chills) from inclusion until fever is absent and the other signs and symptoms reach a score* of 1 or 0.
  *Scores will be classified from 0 to 3, as follows: absent (0), mild (1), moderate (2), or severe (3), according to the Influenza-like Illness Signs and Symptoms Scale (ILISSS).
Evaluation of the Effectiveness of Nitazoxanide in the Outpatient Treatment of Influenza | From enrollment to the end of treatment will last up to 60 days
  The evaluation will be conducted by comparing the nitazoxanide and placebo groups regarding the time to symptom resolution (fever, cough, runny nose, nasal congestion, sore throat, fatigue, headache, muscle pain, sweating, or chills) from inclusion until fever is absent and the other signs and symptoms reach a score* of 1 or 0.
  *Scores will be classified from 0 to 3, as follows: absent (0), mild (1), moderate (2), or severe (3), according to the Influenza-like Illness Signs and Symptoms Scale (ILISSS).

SECONDARY OUTCOMES:
Evaluation of the Effectiveness of Nitazoxanide in the Outpatient Treatment of COVID-19 | From enrollment to the end of treatment will last up to 60 days
  The evaluation will be conducted by comparing the nitazoxanide and placebo groups regarding the time to symptom resolution (fever, cough, runny nose, nasal congestion, sore throat, fatigue, headache, muscle pain, sweating, or chills) from inclusion until fever is absent and the other signs and symptoms reach a score* of 1 or 0, for participants who developed symptoms less than 24 hours before inclusion.
Evaluation of the Effectiveness of Nitazoxanide in the Outpatient Treatment of Influenza | From enrollment to the end of treatment will last up to 60 days
  The evaluation will be conducted by comparing the nitazoxanide and placebo groups regarding the time to symptom resolution (fever, cough, runny nose, nasal congestion, sore throat, fatigue, headache, muscle pain, sweating, or chills) from inclusion until fever is absent and the other signs and symptoms reach a score* of 1 or 0, for participants who developed symptoms less than 24 hours before inclusion.
Evaluation of the Protective Effect of Nitazoxanide on the Development of Cognitive Changes Resulting from COVID-19 | From enrollment to the end of treatment will last up to 60 days
  The evaluation will be conducted by comparing the nitazoxanide and placebo groups regarding cognitive impairments observed between V6 and V8 in the following tests:
  1. MoCA
  2. TMT-A
  3. TMT-B
Evaluation of the Protective Effect of Nitazoxanide on the Development of Pulmonary Dysfunction Resulting from COVID-19 | From enrollment to the end of treatment will last up to 60 days
  The evaluation will be conducted by comparing the nitazoxanide and placebo groups regarding changes in spirometric parameters observed between V6 and V8:
  1. FVC
  2. FEV1
  3. FVC/FEV1
Evaluation of the Effectiveness of Nitazoxanide in Preventing Bacterial Complications | From enrollment to the end of treatment will last up to 60 days
  The evaluation will be conducted by comparing the nitazoxanide and placebo groups regarding the incidence of antibacterial medication prescriptions.
Evaluation of the Effectiveness of Nitazoxanide in Preventing Hospitalization | From enrollment to the end of treatment will last up to 60 days
  The evaluation will be conducted by comparing the nitazoxanide and placebo groups regarding the incidence of hospitalization.
Evaluation of the Safety of Nitazoxanide in Participants with COVID-19 or Influenza Under Outpatient Treatment | From enrollment to the end of treatment will last up to 60 days
  The evaluation will be conducted by comparing the nitazoxanide and placebo groups regarding the incidence and classification of treatment-emergent adverse events in terms of type, frequency, and severity.v